CLINICAL TRIAL: NCT04274738
Title: A Phase 1b Trial of Mavorixafor, an Oral CXCR4 Antagonist, in Combination With Ibrutinib in Patients With Waldenstrom's Macroglobulinemia (WM) Whose Tumors Express Mutations in MYD88 and CXCR4
Brief Title: A Study of Mavorixafor in Combination With Ibrutinib in Participants With Waldenstrom's Macroglobulinemia (WM) Whose Tumors Express Mutations in MYD88 and CXCR4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: X4 Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X4P-001-204; 2019-003909-95 (EudraCT Number)
Record Dates: First submitted 2020-02-12; First posted 2020-02-18 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Waldenstrom's Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — mavorixafor; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mavorixafor and Ibrutinib (Experimental): Each participants will initially receive mavorixafor at Dose Level 1 (200 mg QD) in combination with ibrutinib 420 mg. Cohort A will comprise the first 6 participants enrolled in the study that complete at least their first cycle at Dose Level 2 (400 mg QD). Cohort A participants will start at Dose Level 1 and be allowed to dose escalate after the first cycle to Dose Level 2, if no DLTs are observed during the first cycle of each participant. Cohort B will comprise the next 6 participants enrolled into the study that complete at least their 1st cycle at Dose Level 3 (600 mg QD). Cohort B participants will start at Dose Level 1 and be allowed to dose escalate up to Dose Levels 2 and 3. Cohort C will comprise the remainder of participants enrolled up to the total of 18. Cohort C participants will start at Dose Level 1 and be allowed to escalate to 400 and 600 mg after each dose level has been deemed safe by participants from Cohort A and B.
  Interventions: Drug: Mavorixafor; Drug: Ibrutinib

INTERVENTIONS:
Drug: Mavorixafor — Mavorixafor capsules will be administered per dose and schedule specified in the arm.
  Other Names: X4P-001
Drug: Ibrutinib — Ibrutinib capsules will be administered per dose and schedule specified in the arm.

SUMMARY:
The primary objective of the study is to establish a pharmacologically active dose of mavorixafor in combination with ibrutinib based on pooled safety, clinical response, pharmacokinetic (PK) and pharmacodynamic (PD) data to select the recommended dose for a randomized registrations trial.

DETAILED DESCRIPTION:
This is an intrapatient dose-escalation study. Three dose levels of mavorixafor will be explored: 200 milligrams (mg) once daily (QD) (dose level 1), 400 mg QD (dose level 2), and 600 mg QD (dose level 3). Ibrutinib will be administered at its labeled dose for participants with WM, 420 mg orally QD. Each treatment cycle will be 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to sign informed consent
* Participants must have a clinicopathological diagnosis of WM and must meet the criteria for treatment using consensus panel criteria from the Second International Workshop on Waldenstrom's Macroglobulinemia
* Participant' WM must have confirmed MYD88L265P and CXCR4WHIM mutations
* Participants must have measurable disease, defined as the presence of serum IgM with a minimum IgM level of greater than or equal to (≥) 2 * the upper limit of normal (ULN)
* Participants may be treatment naïve or have received up to 3 prior treatment regimens for WM
* Participants must have an ECOG performance status of 0 or 1
* Participants must meet the following organ and bone marrow requirements:

  i) Absolute neutrophil count greater than (>) 1,000/microliter (μL) ii) Platelet count ≥50,000/μL (platelet transfusion-independent) iii) Hgb ≥8 grams/deciliter (gm/dL) iv) Aspartate aminotransferase and alanine aminotransferase less than or equal to (≤) 2.5 * the ULN and serum total bilirubin ≤1.5 * the ULN, unless secondary to known Gilbert's Syndrome or hepatic infiltration by WM, in which case the total bilirubin must be ≤3 * the ULN and direct bilirubin ≤1.5 × the ULN v) Serum lipase ≤1.5 * the ULN vi) Serum creatinine ≤2 * the ULN or a creatinine clearance of ≥30 milliliters (ml)/minute based on the Cockcroft-Gault equation
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test
* WOCBP who are heterosexually active and male participants with female sexual partners of childbearing potential must agree to use an effective method of contraception (for example; oral contraceptives, double-barrier methods such as a condom and a diaphragm, intrauterine device) during the study and for 4 weeks after the last dose of study medication, or to abstain from sexual intercourse for this time; a woman not of childbearing potential is one who has undergone a bilateral oophorectomy or who is postmenopausal, defined as the absence of menstrual periods for 12 consecutive months
* Participants must be willing and capable of complying with the requirements of the study

Exclusion Criteria:

* Participants with symptomatic hyperviscosity syndrome; participants who undergo plasmapheresis for hyperviscosity may be considered for enrollment once IgM level is under 4,000 mg/dl
* Participants who have known hypersensitivity to mavorixafor or any of its components or to ibrutinib
* Participants who have previously received a CXCR4 inhibitor or a BTK inhibitor
* Participants who are pregnant or breastfeeding
* Participants with an infection requiring intravenous antibiotics or hospitalization at the scheduled time of the first administration of protocol therapy
* Participants with glycated hemoglobin (HbA1c) >6.5%
* Participants with central nervous system (CNS) lymphoma; participants with suspected CNS lymphoma should undergo appropriate diagnostic studies (magnetic resonance imaging, lumbar puncture) before enrollment to determine if CNS lymphoma is present
* Participants with ongoing acute clinical AEs of National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) Grade >1 resulting from prior cancer therapies or participants receive prior chemotherapy within 2 weeks of initial dosing or prior autologous hematopoietic stem cell transplantation (auto-HSCT) within 6 weeks of initial dosing
* Participants with a history of, or positive serologies for, human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection (participants with HBsAb positivity due to a hepatitis B virus [HBV] vaccination are eligible)
* Participants who have had within the past 6 months, the occurrence or persistence of one or more of the following medical conditions that could not be controlled with usual medical care (for example; required emergency care or hospitalization): hypertension, diabetes, unstable angina, seizure disorder, or myocardial infarction
* Participants with clinically significant cardiac disease, including congestive heart failure consistent with New York Heart Association Class 3 or 4; uncontrolled hypertension, clinically significant angina, clinically significant arrythmias including a history of atrial fibrillationin the last 2 years, corrected QT interval using Fridericia formula of >470 milliseconds (msec) or a history of prolonged QT syndrome
* Participants who have had within the past 6 months the occurrence of one or more of the following events: cerebrovascular accident, deep vein thrombosis, pulmonary embolism, hemorrhage (NCI CTCAE Grade 3 or Grade 4), or chronic liver disease (meeting criteria for Child-Pugh Class B or C)
* Participants with prior organ transplantation (prior auto-HSCT are eligible)
* Participants who have an uncontrolled bleeding disorder or require an anticoagulant at the time of study treatment
* Participants with active autoimmune disease requiring systemic steroid administration
* Participants with active second malignancies. (except: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers; any non-hematological malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type)
* Participants who have received an investigational agent within 5 half-lives of the agent; if the half-life of the agent is unknown, participants must wait 4 weeks
* Participants who require strong or moderate inhibitors or inducers of CYP3A4 and potent P-gp inhibitors
* Participants who require medications which are classified as sensitive CYP2D6 substrates
* Participant who have received in the 2 weeks preceding the first dose of protocol treatment, any of the following agents:

  i) Granulocyte colony-stimulating factor or granulocyte-macrophage colony-stimulating factor ii) Systemic corticosteroids in a dose of >10 mg equivalent of prednisone daily; topical, ophthalmic, intranasal, and inhalational corticosteroids are permitted iii) Any other immunomodulating agents, including but not limited to interferon alpha, interleukin (IL)-2, mycophenolate, antibodies to tumor necrosis factor (TNF)-α, soluble TNF receptors, Janus kinase inhibitors, or IL-23 antagonists
* Participants with any other medical, personal, social, or psychiatric condition that, in the opinion of the Investigator, may potentially compromise the safety or compliance of the participant or precludes the participant's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With DLTs | Cycle 1 (28 days)
Percent Change From Baseline in Immunoglobulin M (IgM) at Cycle 1 | Baseline, at the end of Cycle 1 (cycle length = 28 days)
Percent Change From Baseline in IgM at Cycle 2 | Baseline, at the end of Cycle 2 (cycle length = 28 days)
Percent Change From Baseline in IgM at Cycle 3 | Baseline, at the end of Cycle 3 (cycle length = 28 days)
Percent Change From Baseline in Hemoglobin (Hgb) at Cycle 1 | Baseline, at the end of Cycle 1 (cycle length = 28 days)
Percent Change From Baseline in Hgb at Cycle 2 | Baseline, at the end of Cycle 2 (cycle length = 28 days)
Percent Change From Baseline in Hgb at Cycle 3 | Baseline, at the end of Cycle 3 (cycle length = 28 days)
Maximum Observed Plasma Concentration (Cmax) of Mavorixafor | Pre-dose, 0.5, 1, 2, 4, 6, and 8 to 10 hours post-dose on Day 1 and Day 21 of Cycle 1, 2, and 3 (each cycle length = 28 days)
Cmax of Ibrutinib | Pre-dose, 0.5, 1, 2, 4, 6, and 8 to 10 hours post-dose on Day 1 and Day 21 of Cycle 1, 2, and 3 (each cycle length = 28 days)
Time to Reach Cmax (Tmax) of Mavorixafor | Pre-dose, 0.5, 1, 2, 4, 6, and 8 to 10 hours post-dose on Day 1 and Day 21 of Cycle 1, 2, and 3 (each cycle length = 28 days)
Tmax of Ibrutinib | Pre-dose, 0.5, 1, 2, 4, 6, and 8 to 10 hours post-dose on Day 1 and Day 21 of Cycle 1, 2, and 3 (each cycle length = 28 days)
Half-Life (t1/2) of Mavorixafor | Pre-dose, 0.5, 1, 2, 4, 6, and 8 to 10 hours post-dose on Day 1 and Day 21 of Cycle 1, 2, and 3 (each cycle length = 28 days)
t1/2 of Ibrutinib | Pre-dose, 0.5, 1, 2, 4, 6, and 8 to 10 hours post-dose on Day 1 and Day 21 of Cycle 1, 2, and 3 (each cycle length = 28 days)
Accumulation Ratio of Mavorixafor | Pre-dose, 0.5, 1, 2, 4, 6, and 8 to 10 hours post-dose on Day 1 and Day 21 of Cycle 1, 2, and 3 (each cycle length = 28 days)
Accumulation Ratio of Ibrutinib | Pre-dose, 0.5, 1, 2, 4, 6, and 8 to 10 hours post-dose on Day 1 and Day 21 of Cycle 1, 2, and 3 (each cycle length = 28 days)
Area Under the Concentration-Time Curve (AUC) of Mavorixafor | Pre-dose, 0.5, 1, 2, 4, 6, and 8 to 10 hours post-dose on Day 1 and Day 21 of Cycle 1, 2, and 3 (each cycle length = 28 days)
AUC of Ibrutinib | Pre-dose, 0.5, 1, 2, 4, 6, and 8 to 10 hours post-dose on Day 1 and Day 21 of Cycle 1, 2, and 3 (each cycle length = 28 days)
Clearance of Mavorixafor | Pre-dose, 0.5, 1, 2, 4, 6, and 8 to 10 hours post-dose on Day 1 and Day 21 of Cycle 1, 2, and 3 (each cycle length = 28 days)
Clearance of Ibrutinib | Pre-dose, 0.5, 1, 2, 4, 6, and 8 to 10 hours post-dose on Day 1 and Day 21 of Cycle 1, 2, and 3 (each cycle length = 28 days)
Volume of Distribution (Vd) of Mavorixafor | Pre-dose, 0.5, 1, 2, 4, 6, and 8 to 10 hours post-dose on Day 1 and Day 21 of Cycle 1, 2, and 3 (each cycle length = 28 days)
Vd of Ibrutinib | Pre-dose, 0.5, 1, 2, 4, 6, and 8 to 10 hours post-dose on Day 1 and Day 21 of Cycle 1, 2, and 3 (each cycle length = 28 days)
Change From Baseline in AUC of Absolute Neutrophil Count (ANC) at Cycle 1 | Baseline, at the end of Cycle 1 (cycle length = 28 days)
Change From Baseline in AUC of ANC at Cycle 2 | Baseline, at the end of Cycle 2 (cycle length = 28 days)
Change From Baseline in AUC of ANC at Cycle 3 | Baseline, at the end of Cycle 3 (cycle length = 28 days)
Maximal Change From Baseline in ANC Count at Cycle 1 | Baseline, at the end of Cycle 1 (cycle length = 28 days)
Maximal Change From Baseline in ANC Count at Cycle 2 | Baseline, at the end of Cycle 2 (cycle length = 28 days)
Maximal Change From Baseline in ANC Count at Cycle 3 | Baseline, at the end of Cycle 3 (cycle length = 28 days)

SECONDARY OUTCOMES:
Percent Change From Baseline in Serum IgM Levels Over the Time | Baseline, at each cycle throughout the study (up to approximately 2 years) (cycle length = 28 days)
Change From Baseline in Hgb at Over the Time | Baseline, at each cycle throughout the study (up to approximately 2 years) (cycle length = 28 days)
Major Response Rate | From Baseline up to end of study (up to approximately 2 years)
  Major response rate is defined as percentage of participants with complete response + very good partial response + partial response.
Number of Participants With Adverse Events (AEs) | From Baseline up to end of study (up to approximately 2 years)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mass General Hospital Cancer Center, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas
- University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided